CLINICAL TRIAL: NCT01541449
Title: Observational Study Between People That Use Plaquenil and Those Who do Not in Prevention of AMD.
Brief Title: Plaqenil Role in Prevention of Age Related Macular Degeneration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ZIV-0061-11
Record Dates: First submitted 2012-02-02; First posted 2012-03-01 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-01

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD; PLAQUENIL; CNV
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RA patients treated with plaquenil
- Patients who do not use plaquenil

SUMMARY:
The investigators think that there is a connection between the use of plaquenil and the prevention of Age related macular degeneration (AMD). The investigators believe that the use of plaquenil makes bruch's membrane thicker, thereby preventing Chroidal Neovascularization (CNV) growth.

DETAILED DESCRIPTION:
the study is done by comparing to groups RA patients who take plaquenil Vs. group of patients who do not take plaquenil. after measuring the retina thickness we compare the avg. thickness of both groups.

ELIGIBILITY:
Inclusion Criteria:

* all people who suffer from rheumatoid arthritis (RA) and use plaquenil

Exclusion Criteria:

* patients who did not complete follow-up

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ziv Medical center retina clinic population
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Study Completion 2012-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph pikkel, M.D, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv Medical Center, Safed, Israel